CLINICAL TRIAL: NCT05312502
Title: Effect of Using a Birth Ball on Birth Satisfaction and Pain in Pregnant Women During Labor: A Randomized Controlled Trial
Brief Title: Effect of Using a Birth Ball on Birth Satisfaction and Pain in Pregnant Women During Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Yasemin ERKAL AKSOY, Asistant Prof. Dr., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0000-0002
Record Dates: First submitted 2022-03-21; First posted 2022-04-05 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Pain; Labor Pain; Satisfaction
Keywords: Birth ball; birth satisfaction; pain; midwifery care
MeSH Terms: conditions — Pain; Labor Pain; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: The sample size was 106 pregnant women, 53 in each group, with a known score using the G*Power 3.1.7 program (intervention group=29.19±5.86-control group=26.51±5.13) with 85% power, 0.48 effect size and 0.15 error. was calculated as. Considering data loss, it is planned to reach 10% more pregnant women. Intervention group=57, control group=54 pregnants, and the study was terminated. The women were divided into two groups using the random numbers table in the simple random sampling method. Single blinding was performed on the women participating in the study. However, in order to prevent bias, the researcher who collected the data gave codes to the questionnaire forms of the pregnant women.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Birth Ball (Experimental): In the second stage, the birth ball application was made and followed. Pregnant women with a vaginal opening of 4 cm admitted to the delivery room were instructed to sit on the delivery ball for a total of 30 minutes. A stopwatch clock was used to determine these 30 minutes. The pregnant woman was not asked to sit on the ball all the time, and she could take a break for rest or other needs. The birth ball, which is suitable for women's use, was preferred in 45 cm dimensions, and the pilates circle was used as a stabilizer. Under the supervision of the researcher, the pregnant women sat upright on the ball and began to rock back and forth. Meanwhile, the researcher held the pregnant woman's hand. In order for the pregnant woman not to lose her balance, the birth ball was placed on a pilates circle and she was supported by the researcher in making the movements.
  Interventions: Other: Birth Ball
- Control (No Intervention): A routine care was performed.

INTERVENTIONS:
Other: Birth Ball — During labour, the pregnant woman was positioned using a birth ball.
  Arms: Experimental: Birth Ball

SUMMARY:
H0: There is no difference between birth satisfaction and pain levels of pregnant women who used and did not use a birth ball during labor.

H1: There is a difference between birth satisfaction and pain levels of pregnant women who used and did not use a birth ball during the birth process.

ELIGIBILITY:
Inclusion Criteria:

* the consent of the pregnant women to participate in the study,
* have signed the informed consent form,
* be over the age of 18,
* Vaginal opening was determined as 4 cm

Exclusion Criteria:

* Having a psychologically diagnosed disorder
* Pregnant women diagnosed with risky pregnancy

Ages: 19 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 111 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Introductory Information Form | pre-intervention
  The form consisting of 13 questions was prepared by the researcher in order to describe the sociodemographic characteristics and current health status of women.
Birth Process Follow-up Form | during the intervention
  It was created by the researcher in order to obtain information about the progress of birth and the characteristics of the fetus during the birth process of the pregnant. In the form, there are questions including the hour and subsequent follow-up hours when the vaginal opening is 4 cm, dilatation, fetal heartbeat, whether there is oxytocin administration, the duration and frequency of contractions, and the characteristics of the amniotic fluid.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | during the intervention
  It is a measurement usually used to evaluate pain from 0 (no pain) to 10 (unbearable pain). A 10 cm vertical form was used in the study. Pain level was evaluated with VAS during each follow-up of the pregnant woman.
Birth Satisfaction Scale-Short Form (DME-F) | in the first hour in postpartum period
  The short form of the scale was revised by Martin et al. in 2016 to evaluate the birth satisfaction levels of women (Martin et al., 2016). The Turkish validity and reliability study was conducted by Serhatlıoğlu et al. in 2018 (Göncü Serhatlıoğlu et al., 2018). The scale consists of 10 items and a minimum of 0 and a maximum of 40 points can be obtained. The items of the scale are in a 5-point Likert type and are scored as Strongly agree (4 points)-Strongly Disagree (0 points).

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Ali Kemal Belviranlı Gynecology and Pediatrics Hospital, Konya, Turkey (Türkiye)

REFERENCES:
- [Derived] Kilic S, Dereli Yilmaz S. Virtual Reality Headset Simulating a Nature Environment to Improve Health Outcomes in Pregnant Women: A Randomized-Controlled Trial. Clin Nurs Res. 2023 Nov;32(8):1104-1114. doi: 10.1177/10547738231184923. Epub 2023 Jul 5. PMID 37408298